CLINICAL TRIAL: NCT02231931
Title: Relative Bioavailability of a Single Oral Dose of Digoxin, Furosemide, Metformin, and Rosuvastatin Given Alone and All Together as a Cocktail, and Investigation of the Effect of Increased Doses of Metformin or Furosemide on Relative Bioavailability of the Other Cocktail Compounds in Healthy Male Subjects
Brief Title: Drug-drug Interaction Between Digoxin, Furosemide, Metformin, and Rosuvastatin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 352.2082; 2014-001940-40 (EudraCT Number: EudraCT)
Record Dates: First submitted 2014-09-03; First posted 2014-09-04 (Estimated); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Healthy
MeSH Terms: interventions — Digoxin; Rosuvastatin Calcium; Furosemide; Metformin

ARMS (7):
- A (Reference 1) Digoxin (Experimental): 1 tablet as single dose, fasted
  Interventions: Drug: Digoxin
- B (Reference 2) Furosemide (Experimental): oral solution, as single dose, fasted
  Interventions: Drug: Furosemide
- C (Reference 3) Metformin hydrochloride (Experimental): 1 film-coated tablet as single dose, fasted
  Interventions: Drug: Metformin hydrochloride
- D (Reference 4) Rosuvastatin (Experimental): 1 film-coated tablet as single dose, fasted
  Interventions: Drug: Rosuvastatin
- E (Test) 1 (Experimental): Digoxin (1 tablet), Furosemide (0.5 mL oral solution), Metformin hydrochloride (1 film-coated tablet), Rosuvastatin (1 film-coated tablet), fasted
  Interventions: Drug: Digoxin, Furosemide, Metformin hydrochloride, Rosuvastatin
- F (Test 2) (Experimental): Digoxin (1 tablet), Furosemide (0.5 mL oral solution), Metformin hydrochloride (2 film-coated tablets), Rosuvastatin (1 film-coated tablet), fasted
  Interventions: Drug: Digoxin, Furosemide, Metformin hydrochloride, Rosuvastatin
- G (Test 3) (Experimental): Digoxin (1 tablet), Furosemide (2.0 mL oral solution), Metformin hydrochloride (1 film-coated tablet), Rosuvastatin (1 film-coated tablet), fasted
  Interventions: Drug: Digoxin, Furosemide, Metformin hydrochloride, Rosuvastatin

INTERVENTIONS:
Drug: Digoxin — single dose, fasted
  Arms: A (Reference 1) Digoxin
Drug: Rosuvastatin — single dose, fasted
  Arms: D (Reference 4) Rosuvastatin
Drug: Digoxin, Furosemide, Metformin hydrochloride, Rosuvastatin — fasted
  Arms: E (Test) 1
Drug: Digoxin, Furosemide, Metformin hydrochloride, Rosuvastatin — fasted
  Arms: G (Test 3)
Drug: Metformin hydrochloride — single dose, fasted
  Arms: C (Reference 3) Metformin hydrochloride
Drug: Digoxin, Furosemide, Metformin hydrochloride, Rosuvastatin — fasted
  Arms: F (Test 2)
Drug: Furosemide — single dose, fasted
  Arms: B (Reference 2) Furosemide

SUMMARY:
To investigate the mutual interaction potential of digoxin, furosemide, metformin, and rosuvastatin when given alone or together as a cocktail, and to investigate the effect of high doses of metformin or furosemide on pharmacokinetics of the other cocktail compounds

ELIGIBILITY:
Inclusion criteria:

1. Healthy male subjects according to the investigator´s assessment, based on a complete medical history including a physical examination, vital signs (Blood Pressure, Pulse Rate), 12-lead Electrocardiogram, and clinical laboratory tests
2. Age of 18 to 50 years (incl.)
3. Body Mass Index of 18.5 to 29.9 kg/m2 (incl.)
4. Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and local legislation

Exclusion criteria:

1. Any finding in the medical examination (including Blood Pressure, Pulse Rate, or Electrocardiogram) is deviating from normal and judged as clinically relevant by the investigator
2. Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 bpm
3. Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
4. Any evidence of a concomitant disease judged as clinically relevant by the investigator
5. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological, or hormonal disorders
6. Surgery of the gastrointestinal tract that could interfere with kinetics of the trial medication (except appendectomy and simple hernia repair)
7. Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2015-01-01 (Actual); Study Completion 2015-01-01 (Actual)

PRIMARY OUTCOMES:
Digoxin, Metformin, Rosuvastatin: AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point) | up to 96 hours
Furosemide: AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point) | up to 36 hours
Furosemide: Cmax (maximum measured concentration of the analyte in plasma) | up to 36 hours
Digoxin, Metformin, Rosuvastatin: Cmax (maximum measured concentration of the analyte in plasma) | up to 96 hours

SECONDARY OUTCOMES:
Furosemide: AUC0-inf (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | up to 36 hours
Digoxin, Metformin, Rosuvastatin: AUC0-inf (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | up to 96 hours

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 352.2082.1 Boehringer Ingelheim Investigational Site, Biberach, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency